CLINICAL TRIAL: NCT06431308
Title: Adjuvant Nutritional Therapy to Incretin-based Anti-obesity Medications in the Management of Gastrointestinal Adverse Events During the Up-titration Phase
Brief Title: Nutritional Therapy to Incretin-based Anti-obesity Medications in the Management of Gastrointestinal Adverse Events
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ariel University (Other)
Responsible Party: Principal Investigator, Shiri Sherf Dagan, Principal Investigator, Ariel University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ASMC-0003-24
Record Dates: First submitted 2024-03-28; First posted 2024-05-28 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Obesity; Drug
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional intervention group (Experimental): Nutrition guidance before AOM treatment by registered dietitian (RD) followed by nutrition and behavioral recommendations according to reported gastrointestinal symptom(s).
  Interventions: Behavioral: nutritional intervention
- Control group (No Intervention): * Usual nutrition care treatment for patients treated with Wegovy© or Mounjaro© (RCT).
  * Prior to the initiation of AOM treatment, participant will receive general nutrition guidance based on national recommendations according to the Mediterranean diet.

INTERVENTIONS:
Behavioral: nutritional intervention — A nutrition guidance before initiation of AOM treatment include recommendations for food choices and eating habits to minimize the occurrence and severity of GI symptoms during the up-titration phase, will be given by registered dietitian (RD) from the study team. Next, each week, participants will provide weekly reports of GI symptoms occurrence and severity, by responding to queries sent via WhatsApp/SMS and for occurring symptoms, an automatically structured nutrition and behavioral treatment recommendations will be sent . If participants expressed an interest in personalized dietary guidance on this matter, the study team RD will contact him/her by telephone, within a range of 48 hours, to provide individualized recommendations. Three days after each report of GI symptom(s), participants will receive an additional message and will be asked to report the occurrence and severity of the GI symptom, and their compliance with the specific dietary instructions received.
  Arms: Nutritional intervention group

SUMMARY:
The goal of the study is to evaluate the effect of nutrition intervention on gastrointestinal symptoms, treatment discontinuation rate, nutritional parameters (e.g., dietary intake and eating habits), anthropometric measures, functional parameters, and QOL during the initiation and up-titration phase of incretin-based Anti Obesity Medications (AOM) treatment in patients with overweight/obesity.

The nutrition intervention protocol will be developed based on literature review, focus groups with health care professionals, and patient interviews.

A single-center pilot study will be performed at the Tel-Aviv Assuta Medical Center, among 10 patients who are about to initiate long-term weight management treatment with Wegovy© (semaglutide 2.4 mg), followed by a multi-center, parallel design open-label, RCT, which will be conducted at the Tel-Aviv Assuta Medical Center and Rabin Medical Center - Beilinson Hospital, in 120 patients who are about to initiate long-term weight management treatment with Wegovy© or Mounjaro© .

The intervention group will receive nutrition guidance before AOM treatment by registered dietitian (RD) followed by nutrition and behavioral recommendations according to reported gastrointestinal symptom(s). The control group will receive the usual nutrition care for patients treated with AOM.

Primary outcomes (gastrointestinal symptom assessment) and secondary outcomes (incretin-based AOM discontinuation rate, nutritional parameters, anthropometrics, functional parameters and QOL) will be evaluated by interviews, questionnaires and measurements at baseline, at the end of Wegovy© or Mounjaro© titration phase [20 weeks (T1)] and weekly during the study period (for GI symptoms assessment).

ELIGIBILITY:
Inclusion Criteria:

* individuals aged ≥ 18 years
* eligible to receive AOM [i.e., BMI ≥ 30 kg/m2 or ≥ 27 kg/m2 with at least one adiposity-related coexisting condition (e.g., diabetes or pre-diabetes, hypertension, dyslipidemia, obstructive sleep apnea, fatty liver, cardiovascular disease)]
* who can read and speak Hebrew.

Exclusion Criteria:

* Contraindications or precautious for treatment with Wegovy© or Mounjaro© [i.e., personal or family history of medullary thyroid cancer (MTC), personal history of multiple endocrine neoplasia type 2 (MEN2) syndrome, attempting conception, current pregnancy or breastfeeding]
* previous bariatric surgery or endo-bariatric procedure
* presence of chronic pancreatitis
* treatment with AOM within a month before enrollment
* patients with type 1 diabetes mellitus
* patients who underwent other major GI surgery prior to medication treatment
* patient with underlying GI disease [e.g., gastroparesis, celiac, Inflammatory Bowel Disease (IBD)]
* a positive diagnosis of small-intestinal bacterial overgrowth (SIBO)
* patients with active gastritis, gastroenteritis
* chronic usage of promotility drugs or laxatives
* patients with uncontrolled mental illness
* significant cognitive deterioration
* alcohol consumption exceeding 1 drink per day for women and 2 drinks per day for men .

In addition, participants who decide not to initiate or stop Wegovy© or Mounjaro© treatment for more than two consecutive injections for any reason or who undergo bariatric surgery or endoscopic sleeve gastroplasty during the study period will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal symptoms assessment | Baseline and at the end of the study period (20 weeks)
  GI symptoms rating scale (GSRS) - assess the degree of specific GI complaints Every question is rated by seven graded Likert-type scale (1 represents the absence of troublesome symptoms and 7 represents very troublesome symptoms) while a higher score of the whole questionnaire and by dimension represents more severe symptoms.
Defecation texture | Baseline and at the end of the study period (20 weeks)
  Bristol stool scale - classifying the form of human feces into seven categories. Type 1-2 are considered abnormal hard stools and indicative of constipation type, and type 5-7 are considered abnormally loose/liquid stools and indicative of diarrhea or urgency
Bowel Movement (BM) frequency | Baseline and at the end of the study period (20 weeks)
  will be assessed according to five acceptable categories: >3 BMs/day, 2-3 BMs/day, 1-2 BMs/day, 3-4 BMs/week, <3 BMs/week
Participants gastrointestinal symptoms report | Baseline, at the end of the study period (20 weeks) and weekly until 20 weeks (for subjective GI symptoms report only)
  Participant subjective and objective reporting of GI symptoms

SECONDARY OUTCOMES:
Incretin-based AOM treatment discontinuation rate | At the end of the study period (20 weeks) and weekly until 20 weeks
Anthropometric measures - weight | Change from baseline at the end of the study period (20 weeks)
  Weight (kg) by digital scale
Anthropometric measures - waist circumference (WC) | Change from baseline at the end of the study period (20 weeks)
  will be measured by tape measure (cm)
Body composition - fat mass (kg) | Change from baseline at the end of the study period (20 weeks)
  Body composition analysis using Inbody370S®
Dietary intake | Change from baseline at the end of the study period (20 weeks)
  24-hour dietary recall (24HR)
Eating habits assessment | Change from baseline at the end of the study period (20 weeks)
  General questions regarding eating patterns, hydration and foods intolerance
Eating habits assessment - Control of Eating | Change from baseline at the end of the study period (20 weeks)
  Control of Eating Questionnaire (CoEQ) - The of CoEQ consists of 21 items (19 questions are rated by 100 mm VAS, and two question are open-ended). Greater score represents greater levels of Craving Control.
Functional parameters - muscle strength | Change from baseline at the end of the study period (20 weeks)
  Handgrip (HG) muscle Strength - measure static muscle strength (kg) of the upper extremities by a digital hand dynamometer (Jamar plus digital©)
Functional parameters- leg strength and endurance | Change from baseline at the end of the study period (20 weeks)
  30-seconds sit and stand test - counts the number of times the patient stands in 30 seconds. Higher scores means a better outcome.
Quality of life assessment | Change from baseline at the end of the study period (20 weeks)
  EQ-5D-3L questionnaire -include the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS) .The EQ-5D-3L descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems.The EQ VAS records the patient's self-rated health. Participants will be asked to subjectively rate their overall state of health by using a 0 to 100 VAS, with a higher score reflects a better outcome.
Eating habits assessment - Food preferences | Change from baseline at the end of the study period (20 weeks)
  Leeds Food Preference Questionnaire (LFPQ). The questionnaire involves an explicit evaluation of "liking" and "wanting" for 16 food items that can be categorized as high-fat savory (HFSA), low-fat savory (LFSA), high-fat sweet (HFSW) and low-fat sweet (LFSW). Each food image is scored on a 100-mm VAS, while a higher score indicates a stronger preference for that food category. The second sub-task evaluates "implicit wanting" and requires rapid choice between 96 paired combinations of the food images from different categories
Anthropometric measures - height (cm) | Change from baseline at the end of the study period (20 weeks)
  (cm) by altimeter
Body composition- percentage of body fat (BF%) | Change from baseline at the end of the study period (20 weeks)
  Body composition analysis using Inbody370S®
Body composition - fat-free mass (kg) | Change from baseline at the end of the study period (20 weeks)
  Body composition analysis using Inbody370S®
Body composition - skeletal muscle mass (kg) | Change from baseline at the end of the study period (20 weeks)
  Body composition analysis using Inbody370S®

OTHER OUTCOMES:
Biochemical tests | At baseline
  Participants will be asked to provide at T0 biochemical tests obtained during the last 3 months, including complete blood count, lipid profile, fasting glucose, HbA1c, iron, transferrin, ferritin, vitamin B12, folate, vitamin D, albumin and total protein
Demographics - age | At baseline
  years
Demographics - marital status | At baseline
  married, single, divorced or widowed
Demographics - education | At baseline
  less than high school, high school graduate, high school diploma, bachelors degree, masters degree, MD or doctoral degree
Demographics - occupation status | At baseline
  employee full time, employee part time, self-employed or other
Health status - Number of participants with coexisting medical conditions and their types | Baseline and at the end of the study period (20 weeks)
  T2DM, prediabetes, dyslipidemia, HTN,sleep apnea, orthopedic problems, GERD, mental disorder or other
Number of participants using regular medications and their types | Baseline and at the end of the study period (20 weeks)
  usual medications
Smoking habits | Baseline and at the end of the study period (20 weeks)
  smoker, former smoker or never
Number of participants using supplementation and their Types | Baseline and at the end of the study period (20 weeks)
  multiviamin, Iron, vitamin D, folic acid, vitamin B12, calcium or other
Lifestyle factors - Sleeping habits | Baseline and at the end of the study period (20 weeks)
  sleeping quality on a scale of 0-3 (0- very good, 1-quite good, 2- quite bad, 3- very bad)
Lifestyle factors - frequency of physical activity | Baseline and at the end of the study period (20 weeks)
  number of exercises per week
Lifestyle factors - duration of physical activity | Baseline and at the end of the study period (20 weeks)
  exercise time in minutes
Lifestyle factors - type of physical activity | Baseline and at the end of the study period (20 weeks)
  aerobic or anaerobic

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - Ariel University, Ariel
  - Rabin Medical Center, Beilinson Hospital, Petah Tikva
  - Assuta Medical Center, Tel Aviv